CLINICAL TRIAL: NCT04474704
Title: Use of Cheetah® Non-invasive Cardiac Monitoring System to Guide Discontinuation of Postpartum Magnesium Sulfate in Women With Severe Preeclampsia: A Pilot Randomized Control Trial
Brief Title: Use of Cheetah® Cardiac Monitoring System to Guide Discontinuation of Magnesium Sulfate in Women With Severe Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Maged Costantine, MD, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020H0264
Record Dates: First submitted 2020-07-08; First posted 2020-07-17 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Preeclampsia With Severe Features
Keywords: preeclampsia with severe features; magnesium sulfate; Systemic Vascular Resistance; non-invasive cardiac monitoring
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cheetah® non-invasive cardiac monitoring system (Experimental): Using the Cheetah® device to aid in an individualized duration of magnesium sulfate based on reduction in Systemic Vascular Resistance (SVR), up to a maximum of 24 hours postpartum.
  Interventions: Device: Cheetah® non-invasive cardiac monitoring system
- Standard of care (Other): 24 hours of postpartum magnesium sulfate (current arbitrary standard of care)
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Cheetah® non-invasive cardiac monitoring system — Cheetah® non-invasive cardiac monitor system will be used to individually determine the duration of magnesium sulfate postpartum (guided by timing of reduction in Systemic Vascular Resistance (SVR))
  Arms: Cheetah® non-invasive cardiac monitoring system
Other: Standard of care — 24 hours of postpartum magnesium sulfate
  Arms: Standard of care

SUMMARY:
This is a single site pilot randomized, controlled, trial randomizing patients with PE with severe features to one of 2 groups:

* 24 hours of postpartum magnesium sulfate (current arbitrary standard of care)
* Using the Cheetah® device to aid in an individualized duration of magnesium sulfate.

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia with severe features, diagnosed using the American Congress of Obstetricians and Gynecologists (ACOG) standard criteria 4 requiring magnesium sulfate
* Females older than 18 years of age
* Singleton pregnancy
* Gestational age greater than 24 0/7 weeks
* The patient is physically and mentally able to understand the informed consent and is willing to participate in this study
* Able to speak English or Spanish

Exclusion Criteria:

* Multiple gestation
* Prisoners
* Patients with chronic renal insufficiency or epilepsy
* Known cardiovascular disease
* Patients with contraindications to magnesium sulfate use (e.g. myasthenia gravis)
* Patients with eclampsia or HELLP syndrome
* Contraindications for magnesium sulfate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maged Costantine, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care
Started | 21 | 26
Completed | 21 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care | Total
Number analyzed (Participants) | 21 | 26 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5.5) | 30 (5.5) | 30.4 (5.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black race | 4 | 6 | 10
  White race | 17 | 20 | 37
  Hispanic ethnicity | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 26 | 47
Nulliparity [Count of Participants; unit: Participants] | 12 | 14 | 26
BMI at delivery [Mean (Standard Deviation); unit: Kg/m2] | 37.3 (7.7) | 39.1 (9.9) | 38.3 (8.9)
Gestational age at delivery [Median (Inter-Quartile Range); unit: weeks] | 36 [33 to 37] | 36 [34 to 38] | 36 [33.5 to 37.5]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Magnesium Sulfate Use in the Postpartum Period Defined as the Duration in Hours Between Delivery and Discontinuation of Magnesium Sulfate.
Time Frame: up to 24 hours postpartum
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care
Number analyzed (Participants) | 21 | 26
hours | 21.6 (4.7) | 24 (0)

2. Secondary Outcome: Composite of Postpartum Adverse Outcomes
Description: any of the following: use of acute anti-hypertensive medications for persistently severe range blood pressure (defined as >160/110 persistent after 15 min), need for more than one dose of acute anti-hypertensive medications, need to restart Mg (for persistent neurological symptoms), postpartum readmission for PE, as well as the development of pulmonary edema, HELLP, or eclampsia
Time Frame: up to 4 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care
Number analyzed (Participants) | 21 | 26
Participants | 6 | 7

3. Secondary Outcome: Evaluating Incidence of Need to Restart Magnesium Sulfate
Time Frame: up to 1 week postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care
Number analyzed (Participants) | 21 | 26
Participants | 0 | 0

4. Secondary Outcome: Evaluating Number of Participants With Hospital Readmission for Preeclampsia
Time Frame: up to 4 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care
Number analyzed (Participants) | 21 | 26
Participants | 0 | 1

5. Secondary Outcome: Use of Acute Anti-hypertensive Medications
Time Frame: Up to 5 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care
Number analyzed (Participants) | 21 | 26
Participants | 6 | 7

6. Secondary Outcome: Need for More Than 1 Dose of Anti-hypertensive Medication
Time Frame: Up to 5 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care
Number analyzed (Participants) | 21 | 26
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: After up to 4 weeks postpartum
Arm/Group | Cheetah® Non-invasive Cardiac Monitoring System | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/26
Other Adverse Events (participants affected / at risk) | 0/21 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/04/NCT04474704/Prot_SAP_000.pdf